CLINICAL TRIAL: NCT03356873
Title: Impact of Correction of Vitamin D Deficiency in Oxidative Stress in Patients With Impaired Glucose Tolerance: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Impact of Correction of Vitamin D Deficiency in Oxidative Stress in Patients With Prediabetes (VICOX)
Acronym: VICOX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID19
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIA-981-13/14-1
Record Dates: First submitted 2017-10-20; First posted 2017-11-29 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Vitamin D Deficiency; Glucose Intolerance; Oxidative Stress; Insulin Resistance
MeSH Terms: conditions — Vitamin D Deficiency; Glucose Intolerance; Insulin Resistance | interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Vitamin D 5000 units capsules, 20 capsules per week during four weeks (total 400,000 units)
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): Identical placebo capsules, 20 capsules per week during four weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin D — Vitamin D supplementation
  Other Names: Vitamin D3
  Arms: Active
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The investigators aim to determine the effect of the correction of vitamin D in vitamin D deficient patients (<15ng/ml) in oxidative stress and insulin resistance in patients with impaired glucose tolerance. Vitamin D deficiency has been associated with chronic low-grade inflammation, diabetes mellitus type 2, cardiovascular risk and increased prevalence of coronary heart disease, cerebrovascular disease and myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Women, 18 to 70 years, glucose intolerance (post-2 hour 75-grams glucose load > or equal 140 mg/dl), 25-hydroxy vitamin D concentration < or equal 15 ng/ml

Exclusion Criteria:

* Diabetes, systemic inflammatory disorders, treatment with statins, metformin or fibrates, renal insufficiency, intestinal malabsorption

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

PRIMARY OUTCOMES:
Change in anti-oxidant capacity measured in serum | One month
  Change in serum anti-oxidant capacity after one month

SECONDARY OUTCOMES:
Change in homeostasis model assessment (HOMA) index measured in serum | One month
  Change in homeostasis model assessment (HOMA) index after one month

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico